CLINICAL TRIAL: NCT02159885
Title: Telemedici ne Management of Veterans With Newly Diagnosed Obstructiv e Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01473
Record Dates: First submitted 2014-04-28; First posted 2014-06-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; adherence; telemedicine; auto-titrating continuous positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring (Experimental): In this arm, subjects will receive usual care at the sleep clinic as well as telemonitoring of their use of their automatically adjusting continuous positive airway pressure pressure (APAP) machine. They will receiving phone calls for poor adherence and/or poor efficacy of treatment.
  Interventions: Other: Telemonitoring
- Usual Care (No Intervention): Subjects in this arm will receive "usual care" for management of obstructive sleep apnea and use of automatically titrating continuous positive airway pressure.

INTERVENTIONS:
Other: Telemonitoring
  Arms: Telemonitoring

SUMMARY:
Automatically titrating continuous positive airway pressure (APAP) and continuous positive airway pressure (CPAP) are considered first-line treatments for obstructive sleep apnea. There is a growing body of evidence that suggests that early patient education and intervention may improve adherence with positive airway pressure. The investigators plan a prospective, randomized trial to see if telemonitoring in the first several weeks of PAP therapy improves adherence following 3 months of treatment.

DETAILED DESCRIPTION:
Obstructive sleep apnea is a high-priority clinical condition for the Veterans Health Administration. With approximately 2% of middle-aged women and 4% of middle-aged men having OSA, the disorder places significant burden on the healthcare system. Obstructive sleep apnea (OSA) has been linked to major cardiovascular disorders such as coronary artery disease, congestive heart failure, hypertension, and stroke, as well as increased risk for motor vehicle crashes. Positive airway pressure (PAP) therapy is considered the treatment of choice for obstructive sleep apnea. However, adherence rates with CPAP and APAP therapy are disappointingly low. Veterans, especially those who are socioeconomically disadvantaged and those with psychiatric disease, demonstrate poor adherence when compared to the general population. Effective interventions are needed to improve adherence among patients diagnosed with OSA.

Currently, veterans diagnosed with OSA at the Philadelphia VA sleep center are treated with a home APAP machine that records their adherence on a smart card. They are scheduled for a follow-up appointment within one to three months after their initiation of APAP therapy to discuss questions and concerns regarding the machine as well as the mask and to download their adherence data. Given the limited availability of clinic appointments, some patients may have to wait longer than this.

More recently, APAP machines now distributed through the VA system offer the possibility of using wireless transmissions to track adherence data, including hours of use, mask leak, and apnea-hypopnea index (this transmission does not require hook up to the telephone and does not require the patient to have internet access). This offers the opportunity to see if remote monitoring within the first several weeks of APAP treatment improves adherence, and in turn, improves clinical response to treatment. At the present time, all patients enrolled at Philadelphia Veterans Administration Medical Center (PVAMC) who are newly diagnosed with OSA are being provided with APAP machines with modems that allow for wireless transmissions of data through the Phillips Respironics HIPPA compliant website, www.encoreanywhere.com. Review of the modem data is being performed on a limited basis in some patients. If remote monitoring improves adherence, the investigators may want to implement it for all APAP users. At present, the investigators do not know if this is a clinically effective or cost effective model for delivering health care.

The investigators will have a baseline chart review. It will include assessment of APAP settings (auto-titrate pressure ranges), model and size of mask interface, baseline sleep study results (mean AHI), and review of surveys now obtained as part of routine clinical care at the investigators sleep center, including: Epworth Sleepiness Scale (ESS) score, functional outcomes of sleep questionnaire (FOSQ) score, center for epidemiological studies of depression scale (CES-D score), short form health survey (SF-12), a health survey score and client satisfaction questionnaire (CSQ-8).

Sleep center staff will also perform a chart review to obtain demographic information (age, sex, race), BMI, daytime oxygen saturation (if available), and co-morbidities (congestive heart failure, diabetes, hypertension, obesity, chronic obstructive pulmonary disease (COPD), and depression or other psychological disorders) as part of their problem list in the computerized VA medical record. the investigators will use this chart review to compute a Charlson Morbidity Index.

The investigators then plan to randomize 126 patients to either usual care or usual care in addition to telemonitoring.

Standard of Care Arm: Patients assigned to receive standard of care will be set-up with an APAP machine through Eagle Home Medical, our contracted local home health care agency. Patients will also receive the sleep staff's phone number should they encounter problems with the use of their new equipment. Patients will be scheduled to see a sleep practitioner within one to three months of the initiation of APAP therapy.

At the follow-up office visit, practitioners will assess mask leak, mean daily APAP usage, AHI through either secure digital (SD) cards or Encore Anywhere. Practitioners will also calculate the patient's ESS score and inquire about frequent complications associated with APAP-usage, such as dry mouth and mask discomfort.

After three months of treatment, all patients in the usual care arm will also have their EncoreAnywhere data reviewed. They will receive a phone call from our sleep center staff to assess their experience with their APAP machines. If patients have not had a follow-up clinic visit, they will be scheduled for one. In addition, all subjects will be mailed survey to reassess their functional outcomes including: ESS score, FOSQ- 10, another subjective measurement of sleepiness, the CES-D score, an assessment of depression symptoms, the CSQ-8, an assessment of patient satisfaction, and the SF-12 health survey, an assessment of health.

Telemonitoring Arm: Patients will be set-up with an APAP machine through Eagle Home Medical, our contracted local home health care agency. Patients will also receive the sleep staff's phone number should they encounter problems with the use of their new equipment. Patients will be scheduled to see a sleep practitioner within one to three months of the initiation of APAP therapy. At that follow-up appointment, APAP settings, APAP adherence, mask comfort, humidifier usage, and ESS score will be assessed.

In addition, patients in the telemonitoring arm will have their adherence data monitored by sleep research staff. Patients who demonstrate poor adherence will receive phone calls at scheduled intervals (Day 2, Day 9, and Day 16). Poor adherence is defined as a large mask leak for 30% of the night, 30% or more of days with less than 4 hours of use, or an AHI > 10 events/hr.

Day 2 (Can call up to 120 hours after initiation of treatment) Two days after initiation of APAP data, intervention arm patients will have their data reviewed by the sleep study staff. Patients will receive a follow-up call if any of the following are present: large mask leak, 30% or more of days with less than 4 hours of use, or machine measured average AHI > 10 events/hr. Patients will be assessed for symptoms such as dry mouth, mask issues, or discomfort with the device, or any other problems. Interventions to improve adherence (i.e.: a different mask, chin strap, modifications of pressure settings, modifications of humidifier settings, saline nasal sprays) will then be prescribed if needed. Patients will also be given the sleep center number if they have questions regarding the use of their equipment.

Day 9: (Can call up to 120 hours after Day 9) Patients in the intervention arm will have their data reviewed again. They will receive a follow-up call if poor adherence is noted. Symptoms will be assessed and interventions to improve adherence will be offered.

Day 16: (Can call up to120 hours after Day 16) Patients in the intervention are will have their data reviewed again and called if poor adherence and/or efficacy is noted. Symptoms will be assessed and interventions to improve adherence will be offered.

Three Month Follow-up: All patients will have their EncoreAnywhere data reviewed. If patients have not had a follow-up visit within one to three months of APAP set-up, they will be scheduled for one. Surveys will be mailed to all subjects to reassess functional outcomes, including: ESS, FOSQ, CES-D, SF-12 health survey, and CSQ-8.

ELIGIBILITY:
Inclusion Criteria:

* Male and female veterans at least 18 years of age.
* Ability to read and speak English (assessment instruments and therapy will be available only in English).
* AHI> 5 on baseline home sleep study
* Agree to initiate automatically titrating continuous positive airway pressure (APAP) therapy.
* Completion of clinic questionnaires during initial sleep evaluation

Exclusion Criteria:

* Unwilling to provide informed consent.
* Lack of English fluency. This will be determined when potential subjects are contacted by phone. If they are able to understand the oral consent by correctly completing the mini-quiz, English fluency will be established.
* No telephone access
* Patients previously treated with positive airway pressure.
* Patients enrolled in ongoing VA sleep research studies. Currently all patients enrolled in VA sleep research studies already have their charts flagged.
* Patients receiving their sleep care at VA medical centers other than PVAMC, Fort Dix, Gloucester and Victor J. Saracini (Willow Grove).
* Patients initiated on positive airway pressure treatment while in-patients will also be excluded.
* Patients who are set up with APAP machines without modems will also be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Average daily hours of APAP use | 90 days
  Aim 1: The goal of this project is to determine whether telemedicine monitoring of APAP treatment in the first several weeks of treatment improves adherence following 3 months of treatment. Adherence will be measured objectively by the average daily hours of APAP use over 90 days.

SECONDARY OUTCOMES:
Change in FOSQ-10 score | Change in baseline FOSQ-10 score to the FOSQ-10 score assessed at 90 days
  A secondary goal is determine if telemonitoring of APAP treatment improves functional outcomes. We will assess the change in Functional Outcomes Sleep Questionnaire (our primary functional outcome FOSQ- 10), a disease specific quality of life questionnaire.

OTHER OUTCOMES:
Cost of telemonitoring (exploratory) | 90 days
  Aim 3: A third goal (exploratory) is to examine the cost of telemonitoring from both the provider and patient perspective over a 90 day period of time.
Change in ESS score | Change in ESS score from baseline to ESS assessed at day 90 of treatment.
  We will assess the change ESS score- an assessment of sleepiness
Change in CES-D score | Change in baseline CES-D and and CES-D score assessed at 90 days.
  The CES-D is an assessment of depression symptoms.We will assess this as a functional outcome.
The change in the CSQ-8 score | Change from baseline CSQ-8 to CSQ-8 score at 90 days.
  The CSQ-8 is an assessment of patient satisfaction. We will assess this as a functional outcome.
The change in SF-12 health survey score | Change from baseline SF-12 health survey to the SF-12 health survey score at 90 days.
  The SF-12 is an assessment of overall health.We assess the change in score as a functional outcome.
Mean percentage of days used for greater than 4 hours | 1 and 3 months after initiation of APAP therapy
  We will use this as a marker of adherence
No show rate at follow-up sleep clinic | 3 months after initiation of APAP therapy
  We will use this as a marker of overall adherence
Additional time practitioner spends reviewing EncoreAnywhere and calling patients | 3 months after initiation of APAP therapy
  We will use this as part of evaluation of the cost of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kuna, MD, Principal Investigator — Philadelphia VAMC
Locations (1):
- Philadelphia VAMC, Philadelphia, Pennsylvania, United States